CLINICAL TRIAL: NCT00072670
Title: Phase 2 Study of Yondelis in Men With Advanced Prostate Carcinoma
Brief Title: A Phase 2 Study of Trabectedin (Yondelis) in Adult Male Participants With Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR101850; ET-B-025-02
Record Dates: First submitted 2003-11-07; First posted 2003-11-11 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Advanced prostate cancer; Metastatic prostate cancer; Trabectedin; Yondelis; ET-743
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Trabectedin 0.58 milligram per square meter (mg/m^2) (Experimental): Trabectedin will be administered as 3-hour intravenous infusion at dose of 0.58 mg/m^2 weekly on Day 1, 8 and 15 in 28-day cycle and will be continued until disease progression or unacceptable toxicity.
  Interventions: Drug: Trabectedin
- Trabectedin 1.5 mg/m^2 (Experimental): Trabectedin will be administered at dose of 1.5 mg/m^2 as 24-hour infusion every three weeks, and will be continued until disease progression or unacceptable toxicity.
  Interventions: Drug: Trabectedin
- Trabectedin 1.2 mg/m^2 (Experimental): Trabectedin will be administered at dose of 1.2 mg/m^2 as 24-hour infusion every three weeks, and will be continued until disease progression or unacceptable toxicity.
  Interventions: Drug: Trabectedin

INTERVENTIONS:
Drug: Trabectedin — Trabectedin will be administered intravenously as either 0.58 milligram per square meter (mg/m^2) weekly as 3-hour infusion or 1.5 mg/m^2 or 1.2 mg/m^2 every three weeks as 24-hour infusion until disease progression or unacceptable toxicity.
  Other Names: ET-743; Yondelis

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of trabectedin (ET-743) in adult male participants with advanced metastatic (spread of cancer cells from one part of the body to another) prostate cancer.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), non-randomized, multi-center and Phase 2 study in adult male participants with advanced metastatic prostate cancer. The study consists of 3 parts: Screening (consists of 14 days before study commences on Day -1); Treatment (consists of 4-week dosing cycles wherein trabectedin will be administered as intravenously at a dose of either 0.58 milligram per square meter [mg/m^2] weekly 3-hour infusion, or 1.5 mg/m^2 or 1.2 mg/m^2 every three weeks 24-hour infusion); and Follow-up (until survival after the first dose of trabectedin). Participants will discontinue study treatment at disease progression or unacceptable toxicity unless, in the Investigator's opinion, it is deemed that the participants will continue to derive benefit from trabectedin. Efficacy will be evaluated primarily through decline in prostate-specific antigen (substance in blood that is measured to check for prostate cancer) after 72 hours of therapy on Day 1. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Radiographically documented metastatic disease
* Surgical or chemical castration
* Prostate-specific antigen greater than or equal to (>=) 5 nanogram per milliliter (ng/ml)
* Eastern Cooperative Oncology Group performance status of 0, 1, or 2
* Androgen Independent disease

Exclusion Criteria:

* Treatment with chemotherapy or radiation therapy that was terminated at least 4 weeks before study entry
* Treatment with extensive external beam radiation therapy or radionuclide therapy within 6 weeks of study entry (palliative radiation involving less than 20 percent of bone marrow reserves must have been completed at least 4 weeks before study entry)
* Participant not employing adequate contraception
* Other serious illness or medical conditions as : Uncontrolled congestive heart failure or history of myocardial infection or active angina pectoris within six months preceding registration; active infectious process; chronic active liver disease, including chronic Hepatitis B, chronic Hepatitis C, or cirrhosis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2004-01; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Prostate-Specific Antigen (PSA) Response | Day 1 of each cycle until first documented disease progression up to 4 years
  The PSA response will be evaluated according to National Cancer Institute PSA Working Group criterion, which is, greater than or equal to 50 percent decrease in PSA from Baseline after the first dose of study drug, which would be subsequently confirmed by a measurement, that is, at least 4 or more weeks after initial documentation of PSA.

SECONDARY OUTCOMES:
Duration of Prostate-Specific Antigen Response | Day 1 of each cycle until first documented disease progression up to 4 years
  Duration of Prostate-Specific Antigen (PSA) response will be analyzed in all participants for whom a response will be observed. The Duration of a PSA response is the time from a PSA response to PSA progression.
Time to disease progression | Day 1 of each cycle until first documented disease progression up to 4 years
  Time to disease progression is defined as the time period, from initiation of study treatment until documentation of disease progression. If participant will discontinue the study or lost to follow-up without progression or receive further anticancer therapy after study treatment discontinuation in absence of progression, time to progression will be censored at the time of the last PSA evaluation recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Phase 2 Study of Yondelis in Men With Advanced Prostate Carcinoma — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=4518&filename=CR101850_CSR.pdf